CLINICAL TRIAL: NCT03659240
Title: Prebiotic Effects of a Polyphenol-rich Food Product
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Iowa State University (Other)
Responsible Party: Principal Investigator, Wendy S. White, Associate Professor, Iowa State University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 18-303-00
Record Dates: First submitted 2018-09-03; First posted 2018-09-06 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: Dysbiosis
MeSH Terms: conditions — Dysbiosis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cranberry beverage (Experimental)
  Interventions: Other: Cranberry beverage
- Placebo beverage (Placebo Comparator)
  Interventions: Other: Placebo beverage

INTERVENTIONS:
Other: Cranberry beverage — During the intervention period, research participants will consume a cranberry beverage daily.
  Arms: Cranberry beverage
Other: Placebo beverage — During the intervention period, research participants will consume a placebo beverage daily.
  Arms: Placebo beverage

SUMMARY:
The specific aim for this project will be to investigate a cranberry beverage as a means to restore balance in terms of the relative proportions of the various bacteria that inhabit the large intestine.

ELIGIBILITY:
Inclusion Criteria:

* BMI 27-35 kg/m2
* High waist circumference (men >102 cm and women >88 cm)

Exclusion Criteria:

* Cigarette smoking
* Regular intensive exercise
* Pregnancy or lactation
* Chronic diarrhea, constipation, or other gastrointestinal complaint
* Diabetes mellitus, autoimmune disease, or other chronic disease known to alter the gut microbiota
* Use of medications that affect inflammation or the gut microbiota
* Use of prebiotics, probiotics, synbiotics, vitamins, or other dietary supplements known to affect the gut microbiota
* Aversion to cranberries
* Food allergies
* Lactose intolerance
* Vegetarianism

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2018-10-09 (Actual); Primary Completion 2019-02-24 (Actual); Study Completion 2019-02-24 (Actual)

PRIMARY OUTCOMES:
Fecal microbial community composition and structure | Changes in the fecal microbiota will be measured after a 20-day intervention period
  We will investigate if specific bacterial taxa are stimulated by daily consumption of a cranberry beverage.

CONTACTS AND LOCATIONS:
Locations (1):
- Nutrition and Wellness Research Center, Ames, Iowa, United States